CLINICAL TRIAL: NCT01588626
Title: A Phase I, Single Centre, Open Study to Assess the Pharmacokinetics of Oral AZD6140 After Single Dose in Healthy Japanese Male Volunteers
Brief Title: Study to Assess the Pharmacokinetics of AZD6140 After Single Dose in Healthy Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5133C00001
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Healthy volunteer; Japanese males; PK study
MeSH Terms: interventions — Ticagrelor

ARMS (1):
- AZD6140 (Experimental): single administration of 90 mg dose of AZD6140
  Interventions: Drug: AZD6140

INTERVENTIONS:
Drug: AZD6140 — tablet

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of AZD6140 and its active metabolite, safety, tolerability of AZD6140 following single administration in healthy male Japanese volunteers.

DETAILED DESCRIPTION:
A Phase I, Single Centre, Open Study to Assess the Pharmacokinetics of oral AZD6140 after Single Dose in Healthy Japanese Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject aged between 20 to 45 years inclusive
* Body mass index (BMI=weight/height2) between 18.0 to 27.0 kg/m2 inclusive
* Body weight between 50.0 to 85.0 kg inclusive Provision of written informed consent

Exclusion Criteria:

* Clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator, or positive results on screening tests for serum hepatitis B surface antigen and hepatitis C antibody, syphilis and human immu
* Supine blood pressure > 150 mmHg systolic or > 95 mmHg diastolic or supine pulse > 90 beats per minute (after resting for 10 minutes) Personal or family history of bleeding disorders, or reasonable suspicion of vascular malformations, including aneurysms
* Personal or familial predisposition for thrombotic disorders Clinically significant medical history, including psychiatric disorders and severe allergies

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Description of pharmacokinetics for AZD6140 in terms of: Cmax, tmax, t½, AUC(0-t), AUC, CL/F, Vz/F, MRT, and AUC and Cmax ratios of AR-C124910XX to AZD6140, following single administration of 90 mg dose of AZD6140 in healthy Japanese volunteers. | From day 1 (pre-dose) till Day 4 (72h)
  Maximum Concentration (Cmax), Time to reach maximum (peak) plasma concentration (tmax), Terminal plasma half-life (t½), Area under the plasma concentration-time curve from time zero to time t (AUC(0-t)),Area under the plasma concentration-time curve (AUC), Apparent total clearance of the drug from plasma after oral administration (CL/F), Apparent volume of distribution during terminal phase after non-intravenous administration (Vz/F), Mean residence time (MRT), and AUC and Cmax ratios of AR-C124910XX to AZD6140,
Description of pharmacokinetics profile for AR-C124910XX, which is AZD6140 active metabolite, in terms of: Cmax, tmax, t½, AUC(0-t), AUC, CL/F, Vz/F, MRT, and AUC, following single administration of 90 mg dose of AZD6140 in healthy Japanese volunteers. | From day 1 (pre-dose) till Day 4 (72h)

SECONDARY OUTCOMES:
AZD6140 Safety and tolerability profile in terms of: adverse events, vital signs (blood pressure and pulse rate), electrocardiograms (ECGs), laboratory variables | From Day -1 (pre-dose) up to 7-10 days after dose

CONTACTS AND LOCATIONS:
Overall Officials: Hidenori Komori, MD PHD, Study Director — AstraZeneca R&D Japan; Kyoko Matsuguma, Principal Investigator — Kyushu Clinical Pharmacology Research Clinic
Locations (1):
- Research Site, Fukuoka, Fukuoka, Japan